CLINICAL TRIAL: NCT03969472
Title: Effects of Probiotics and Pelvic Floor Muscle Electrophysiologic Therapy on Endometrium Repair in Patients With Intrauterine Adhesion.
Brief Title: Effects of Probiotics and Electrophysiologic Therapy on Endometrium Repair
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: First Affiliated Hospital, Sun Yat-Sen University (Other)
Responsible Party: Principal Investigator, Yuqing Chen, Chief Physician, First Affiliated Hospital, Sun Yat-Sen University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20190529
Record Dates: First submitted 2019-05-29; First posted 2019-05-31 (Actual); Last update posted 2019-05-31 (Actual); Status verified 2019-05

CONDITIONS: Uterine Endometrial Repair
Keywords: probiotic; Electrophysiologic Therapy; uterine endometrial repair; intrauterine adhesion
MeSH Terms: conditions — Gynatresia | interventions — Probiotics

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- probiotic group (Experimental): apply probiotic after surgery
  Interventions: Drug: probiotics
- Electrophysiologic therapy group (Experimental): apply electrophysiologic therapy after surgery without probiotic
  Interventions: Device: Electrophysiologic Therapy
- control (No Intervention): without electrophysiologic therapy and probiotic after surgery

INTERVENTIONS:
Drug: probiotics — apply probiotic after operation
  Arms: probiotic group
Device: Electrophysiologic Therapy — Pelvic floor electrophysiological therapy is used after surgery
  Arms: Electrophysiologic therapy group

SUMMARY:
This study aimed to investigate the effects of probiotics in combination with pelvic floor muscle electrophysiologic therapy on the uterine endometrial repair and reproductive prognosis in patients after surgery for intrauterine adhesion

DETAILED DESCRIPTION:
Post-traumatic repair disorder of endometrium can cause intrauterine adhesions, amenorrhea and infertility, which seriously endanger women's reproductive health. In our previous study, high throughput sequencing of intrauterine microorganisms showed that the content of lactic acid bacteria in the uterine cavity of patients with intrauterine adhesions was significantly lower than that of normal people. Concurrently, our previous studies found that chronic endometritis can aggravate endometrial fibrosis, then affect the repair of endometrial trauma, and increase the recurrence of intrauterine adhesion. Our previous study also suggest that stem cells are beneficial to the repair of endometrium. Studies have shown that lactic acid can inhibit inflammatory response and regulate the proliferation of intestinal stem cells. So can lactic acid also change the microbial environment in uterine cavity to inhibit endometrial inflammation and regulate the proliferation of endometrial stem cells to help repair endometrial wounds? In addition, electrical stimulation can relieve depression and anxiety and play a sedative effect. In recent years, some studies have shown that pelvic floor electrophysiological therapy can improve the intimal blood flow resistance index of thin endometrium. Therefore, whether or not the pelvic floor electrophysiological therapy can repair the endometrium after the intrauterine adhesion. We expect probiotics and electrophysiologic therapy can promote endometrial repair after electrosurgical resection of intrauterine adhesions.

ELIGIBILITY:
Inclusion Criteria:

(1) Preoper- ative AFS score was ≥9; (2) the prior menstrual cycle was regular, and the sex hormone was normal; (3) patients had fertility requirement; (4) male semen examination appeared normal; (5) there were no severe systemic diseases and no contradictions to aspirin, estrogen, and surgery

Exclusion Criteria:

(1) Preoperative AFS score was <9; (2) prior menstrual cycle was irregular and sex hormone was abnormal, or patients had endocrine factors that caused amenorrhea, menstrual reduction, and infertility; (3) patients had no fertility requirement; (4) patients had male factor infertility; (5) patients had contradictions to estrogen and aspirin such as cancers (breast cancer and endometrial cancer), thrombotic diseases, allergy to antipyretic anal- gesics, severe liver injury, hypoprothrombinemia, vitamin K deficiency, hemophilia, thrombocytopenia, and gastric or duodenal ulcer and asthma

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 120 (Estimated)
Dates: Start 2019-05-05 (Actual); Primary Completion 2020-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Endometrial Thickness | Within the first 3 months after surgery
  All Participants in the Mid Menstrual Measured by Color Doppler Ultrasound

SECONDARY OUTCOMES:
Menstruation Pattern of All Participants | Within the first 3 months after surgery
  A method similar to VAS was employed for the evaluation of post-operative menstruation with 0 as amenorrhea and 100 as normal menstruation.
Reduction of American Fertility Society adhesion score at Second-look hysteroscopy of All Participants | Within the first 3 months after surgery
  The severity and extent of intrauterine adhesions were scored according to a classification system recommended by the American Fertility Society (AFS) (1988 version). A score of 1-4 was considered to represent mild adhesions, a score of 5-8 was considered to represent moderate adhesions and a score of 9-12 represented severe adhesions.

CONTACTS AND LOCATIONS:
Overall Officials: Yuqing Chen, MD, Principal Investigator — First Affiliated Hospital, Sun Yat-Sen University
Locations (1):
- First affiliated hospital of SUN Yat-Sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided